CLINICAL TRIAL: NCT06074731
Title: Diagnostic Possibilities in Ophthalmological Diseases Using Swept Source Optical Coherence Tomography
Status: Recruiting | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Matthias Bolz, Head of Ophthalmology and Optometry, Johannes Kepler University of Linz
Other Study IDs: KUK-Ophthalmology-001
Record Dates: First submitted 2019-01-15; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Retinal Disease; Diabetic Retinopathy; Macular Degeneration
MeSH Terms: conditions — Retinal Diseases; Diabetic Retinopathy; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SS-OCT system Plex Elite 9000 — We will use a commercially available SS-OCT system (Plex Elite 9000; Carl Zeiss Meditec).

SUMMARY:
In this pilot study we want to investigate morphological features acquired by the novel image modality and gain information regarding disease pathomechanism, development and future possible influence on disease management for patients affected by those diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 110 years
* Ability to follow instructions during imaging procedure
* Written Informed consent

Exclusion Criteria:

* Dementia
* Inability to follow instructions during imaging procedure
* Patients who do not give informed consent

Ages: 5 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants will be selected by the Department of Ophthalmology at Kepler University Clinic Linz. All patients of the department scheduled for an outgoing appointment with regular examination in the time period of the study can be included in the study. Patients are being examined in the outgoing clinics with standard examinations. Additionally an image using the Zeiss Plex Elite 9000 Swept Source OCT is being performed. Patients of interest for this pilot study are patients with retinal, choroidal, vascular or glaucomatous changes.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Morphological changes using Swept Source Optical Coherence Tomography | through study completion, an average of 1 year
  Morphological changes in retinal diseases provided by Swept Source Optical

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, Prof. Dr., Principal Investigator — Department for Ophthalmology, Kepler University Hospital GmbH, Johannes Kepler University Linz, Altenberger Strasse 69, 4040 Linz, Austria
Locations (1):
- Department for Ophthalmology and Optometry, Kepler University Hospital GmbH, Johannes Kepler University Linz, Altenberger Strasse 69, 4040 Linz, Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No